CLINICAL TRIAL: NCT03375853
Title: Translational Neuroscience: Response Training for Obesity Treatment
Brief Title: Computerized Response Training Obesity Treatment
Acronym: CC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Flinders University (Other); University of Exeter (Other); Radboud University Medical Center (Other); University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK112762
Record Dates: First submitted 2017-05-17; First posted 2017-12-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Hyperphagia; Feeding and Eating Disorders
Keywords: Obesity; Dissonance; Response Training; Eating Disorder; Computer-based Training
MeSH Terms: conditions — Obesity; Hyperphagia; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (Active Comparator): Participants will complete computer based response training tasks that will incorporate pictures of birds, flowers, and mammals. As part of the computer based training, participants will be instructed to respond or inhibit response to certain of these stimuli in order to bring about a change in the participant response to certain stimuli. These tasks will be structured identically to those presented in the experimental condition, only the appearance and context of the stimuli will be different (i.e., non-food versus food items). The computer tasks described above comprise the Generic Response Training Control Intervention.
  Interventions: Behavioral: Generic Response Training Control Intervention
- Experimental Condition (Experimental): Participants will complete computer-based response training tasks that will incorporate pictures of healthy food, unhealthy food, and glasses of water. As part of the computer-based training, participants will be instructed to respond or inhibit responses to certain of these stimuli in order to bring about a change in the participant response to certain stimuli. These tasks will be structured identically to those presented in the control condition, only the appearance and context of the stimuli will be different (i.e., food versus non-food items). The computer tasks described above comprise the Computer Based Response Training Weight Loss Intervention. To optimize the intervention, we narrowed the low-calorie food stimulus set to make a better distinction between high-calorie and low-calorie foods and we changed the filler images (water and furry mammals) in the go/no-go task from 100% "go" to 50% "go" and 50% "no-go" to measure learning of stimulus-specific respond associations.
  Interventions: Behavioral: Computer Based Response Training Weight Loss Intervention

INTERVENTIONS:
Behavioral: Computer Based Response Training Weight Loss Intervention — Participants complete four computer based training tasks each visit, over the course of a few lab visits. Participants then perform weekly booster sessions in a more natural home or community environment over the internet using the same computer based training tasks.
  Arms: Experimental Condition
Behavioral: Generic Response Training Control Intervention — Participants complete four computer based training tasks each visit, over the course of a few lab visits. Participants then perform weekly booster sessions in a more natural home or community environment over the internet using the same computer based training tasks.
  Arms: Control Condition

SUMMARY:
This project will test whether a food response training intervention produces lasting body fat loss, use objective brain imaging to examine the mechanism of effect of this treatment and investigate the generalizability of the training to non-training foods, and examine factors that should amplify intervention effects to provide a test of the intervention theory. This novel treatment represents a bottom-up implicit training intervention that does not rely on executive control, prolonged caloric deprivation, and expensive clinicians to deliver, like behavioral weight loss treatments that have not produced lasting weight loss. If this computer-based response training intervention produces sustained body fat loss in overweight individuals, it could be easily implemented very broadly at almost no expense, addressing a leading public health problem.

DETAILED DESCRIPTION:
Obesity causes 300,000 US deaths yearly, but most treatments do not result in lasting weight loss. People who show greater brain reward and attention region response, and less inhibitory region response, to high-calorie food images/cues show elevated future weight gain, consistent with the theory that overeating results from a strong approach response to high-calorie food cues paired with a weak inhibitory response. This implies that an intervention that reduces reward and attention region response to such food and increases inhibitory control region response should reduce overeating that is rooted in exposure to pervasive food cues. Computer-based response-inhibition training with high-calorie foods has decreased attentional bias for and intake of the training food, increased inhibitory control, and produced weight loss in overweight participants in 3 proof-of-concept trials, with effects persisting through 6-mo follow-up. A pilot trial found that overweight/obese adults who completed a multi-faceted 4-hr response-inhibition training with high-calorie food images and response-facilitation training with low-calorie food images showed reduced fMRI-assessed reward and attention region response to high-calorie training foods and greater body fat loss than controls who completed a rigorous 4-hr generic response-inhibition/response-facilitation training with non-food images (d=.95), producing a 7% reduction in excess body fat over the 4-wk period. The investigators propose to evaluate a refined and extended version of this response-training intervention.

Aim 1: Randomize 180 overweight/obese adults to a 4-wk response training obesity treatment or a generic inhibition training control condition that both include bi-monthly Internet-delivered booster training for a year and a smart phone response training app that can be used when tempted by high-calorie foods, assessing outcomes at pre, post, and at 3-, 6-, and 12-month follow-ups (e.g., % body fat, the primary outcome).

Aim 2: Use fMRI to test whether reduced reward and attention region response, and increased inhibitory region response to high-calorie food images used and not used in the response training mediate the effects of the intervention on fat loss. The investigators will also test whether during training participants show acute reductions in reward and attention region response, and increases in inhibitory response to high-calorie training food images to capture the learning process, assess generalizability of the intervention to food images not used in training, and collect behavioral data on mediators.

Aim 3: Test whether intervention effects will be stronger for those who show less inhibitory control in response to high-calorie food images, a genetic propensity for greater dopamine signaling in reward circuitry, and greater pretest reward and attention region response, and weaker inhibitory region response to high-calorie food images, based on the theory that response training is more efficacious for those with a strong pre-potent approach tendency to high-calorie foods.

During the Covid-19 shelter-at-home order, we will not measure in person only outcomes including BodPod assessments, height and weight measurement for BMI calculation, electrocardiogram (ECG) assessments and fMRI scanning for all participants that have assessments due during this order.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index Between 25 and 35

Exclusion Criteria:

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Body Fat Change | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in participant's body fat percentage

SECONDARY OUTCOMES:
Change in Eating Disorder Symptoms | Baseline, 1 month, 3 months, 6 months, 12 months
  Eating disorder symptoms as measured with the Eating Disorder Diagnostic Interview
Dietary Restraint, Emotional Eating, and External Eating | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Dietary Restraint, Emotional Eating, and External Eating (aggregate score) as measured by the Dutch Eating Behavior Questionnaire
Change in Disinhibited Eating Behavior | Baseline, 1 month, 3 months, 6 months, 12 months
  Chang in Disinhibited Eating as measured by the Three Factor Eating Questionnaire
Change in Eating in the Absence of Hunger Behavior | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Eating When Not Hungry as measured by the Eating in the Absence of Hunger Questionnaire
Change in Food Addiction Behavior | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Problematic eating patterns associated with symptoms of addictive behaviors as measured by the Yale Food Addiction Scale
Change in Physical Activity | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Physical Activity as measured by the Paffenberger Questionnaire
Change in Alcohol Use Behavior | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Substance use frequency (i.e., number of times per day) for alcohol of participants as measured by the Daily Drinking Questionnaire
Change in Substance Use Behavior | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Substance use frequency (i.e., number of times per day) for common recreational drugs of participants as measured by the Daily Drug Taking Questionnaire
Change in Participant Ratings of Unhealthy Food Palatability | Baseline, 1 month
  Change in Participant behavioral response to food pictures, and subjective palatability rating
Change in Participant Ratings of Food Monetary Value | Baseline, 1 month
  Change in Participant behavioral response to food pictures, and willingness to pay given dollar amounts (aggregate score) for the pictured food
Change in Food Craving and Liking Behavior | Baseline, 1 month, 3 months, 6 months, 12 months
  Change Participant food craving behaviors as measured by the Food Craving and Liking Scale
Change in Body Mass Index | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Participant BMI using standard methods of calculation
Change in mean R-Peak Amplitude | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in mean R-Peak Amplitude measured using three-lead ECG using PowerLab 8 Diagnostic Suite
Change in Heart Rate Variability | Baseline, 1 month, 3 months, 6 months, 12 months
  Change in Heart Rate Variability measured using three-lead ECG using PowerLab 8 Diagnostic Suite

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Stanford University
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yokum S, Bohon C, Berkman E, Stice E. Test-retest reliability of functional MRI food receipt, anticipated receipt, and picture tasks. Am J Clin Nutr. 2021 Aug 2;114(2):764-779. doi: 10.1093/ajcn/nqab096. PMID 33851199